CLINICAL TRIAL: NCT02773394
Title: Protocol to Describe the Actual Situation of Hepatitis C Treatment in Brazil
Brief Title: Study to Describe the Actual Situation of Hepatitis C Treatment in Brazil
Acronym: PICTURE
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR107066; TMC435HPC4013 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2016-04-14; First posted 2016-05-16 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C Virus; Observational; Brazil
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Brazilian participants with Hepatitis C virus (HCV) chronic infection who are registered at the Brazilian reference centers and meet all the inclusion criteria and have sufficient information to identify the diagnosis of chronic HCV infection with identification of genotype.

SUMMARY:
The purpose of the study is to describe: 1) the clinical profile, past and current management of participants with hepatitis C in Brazil reference centers; 2) the current situation about demographics characteristics, liver disease progression and clinical outcomes in Brazilian Hepatitis C virus (HCV) participants naive, in treatment and previously exposed to antiviral treatment without sustained virological response (SVR).

DETAILED DESCRIPTION:
This is an observational, non-interventional, cross-sectional, multicenter study to describe demographic characteristics, treatment performed and clinical outcomes of Brazilian participants with HCV chronic infection in about 12 Brazilian reference centers. It will expect that approximately 2000 participants will be enrolled in the study. Analysis set will consist of participants with HCV chronic infection who are registered at the Brazilian reference centers and meet all the inclusion criteria and have sufficient information to identify the diagnosis of chronic HCV infection with identification of genotype. The study related data will be collected from the medical records in the predesigned electronic Case Report Form (eCRF).

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosis confirmed with Hepatitis C infection being followed into the reference centers
* There is no restriction on fibrosis stage or clinical liver disease
* There is no restriction for comorbities or coinfections
* Diagnosis of chronic HCV infection detected by anti-HCV (ELISA assays), HCV Ribonucleic acid (RNA) (polymerase chain reaction [PCR] reaction) with identification of genotype

Exclusion Criteria:

* Male or female participant with age greater than or equal to 18 years
* participating in another interventional clinical trial
* Treated participants who achieved sustained Virological Response (SVR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Analysis set will consist of participants with Hepatitis C virus (HCV) chronic infection who are registered at the Brazilian reference centers and meet all the inclusion criteria and have sufficient information to identify the diagnosis of chronic HCV infection with identification of genotype.
Sampling Method: Non-Probability Sample
Enrollment: 1649 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with chronic hepatitis C infection | Day 1
  Data will be collected through medical records of the participants.
Date of last visit | Day 1
Number of Participants with chronic hepatitis C infection Reported Based on City and States | Day 1
  Data will be collected through medical records of the participants.
Number of Participants with chronic hepatitis C infection Based on precedence | Day 1
  Data will be collected through medical records of the participants.
Mean Age of Participants with chronic hepatitis C infection | Day 1
  Data will be collected through medical records of the participants.
Number of Males and Females with chronic hepatitis C infection | Day 1
  Data will be collected through medical records of the participants.
Number of participants with chronic hepatitis C infection Reported Based on Race | Day 1
  Data will be collected through medical records of the participants.
Mode of Hepatitis C virus (HCV) transmission | Day 1
  Data will be collected through medical records of the participants. Mode of HCV transmission route (unsafe injections, hemodialysis, infection drug use, blood transfusion, sexual transmission, vertical transmission, unknown, other) will be analysed by number of participants infected with HCV per transmission route.
Duration of diagnosis of chronic hepatitis C infection | Day 1
  Data will be collected through medical records of the participants.
HCV genotype and subtype | Day 1
  Data will be collected through medical records of the participants.
Liver characteristics: Number of Participants with extra hepatic manifestations | Day 1
  Data will be collected through medical records of the participants. Presence or absence of extra hepatic manifestations (cryoglobulinemia, lymphoma, Sjogren syndrome, glomerulopathy, Porphyria cutanea tarda, liquen planus, diabetes mellitus, thyroiditis, arthralgia).
Liver characteristics: Number of Participants with presence of comorbidities | Day 1
  Data will be collected through medical records of the participants. Presence of comorbidities (amount of alcohol ingestion, metabolic syndrome, hepatocellular carcinoma, organ transplantation, diabetes, immunodeficiency, renal insufficiency and dialysis, use of drugs) will be collected.
Liver characteristics: Model for End-Stage Liver Disease (MELD) Score and Child Pugh score | Day 1
  MELD is a scoring system for assessing the severity of chronic liver disease. Child-Pugh classification assesses the prognosis of chronic liver disease by 5 clinical measures, scored 1-3 each (most severe derangement=3). Score range: 5 (best prognosis) to 15 (worst prognosis).
Liver characteristics: Number of Participants with Fibrosis based on Fibroscan | Day 1
  Data will be collected through medical records of the participants.
Number of Participants with Coinfections | Day 1
  Data will be collected through medical records of the participants.
HCV treatment status on Day 1: Percentage of participants receiving antiviral treatment | Day 1
  Data will be collected through medical records of the participants.
HCV treatment status on Day 1: Causes of interruption in treatment | Day 1
  Data will be collected through medical records of the participants. Causes of interruption to antiviral therapy will be collected and reported.
HCV treatment status on Day 1: Number of participants treated without Sustained Virological Response (SVR) | Day 1
  Data will be collected through medical records of the participants.
Treatment regimen | Day 1
  The drugs used and time of treatment will be collected through medical records of the participants.
Number of participants with Adverse Events (AEs) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (8):
- Brazil (8):
  - Goiânia
  - Porto Alegre
  - Porto Velho
  - Recife
  - Rio Branco
  - Rio de Janeiro
  - Salvador
  - São Paulo